CLINICAL TRIAL: NCT01015547
Title: Comparison of Anti-TNF Therapy Plus Methotrexate, Combination Therapy of DMARDs, and Methotrexate Alone in Very Early Polyarticular Juvenile Idiopathic Arthritis. A National Randomized Multicenter Clinical Trial.
Brief Title: Aggressive Combination Drug Therapy in Very Early Polyarticular Juvenile Idiopathic Arthritis
Acronym: ACUTE-JIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Foundation for Paediatric Research, Finland (Other); Päivikki and Sakari Sohlberg Foundation, Finland (Other); Rheumatism Foundation Hospital (Other); Scandinavian Rheumatology Research Foundation (Unknown); Paijat-Hame Hospital District (Other)
Responsible Party: Principal Investigator, Pirjo Tynjala, MD PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211864, 318/E0/2002; 211864 (Registry Identifier: www.hus.fi)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: juvenile idiopathic arthritis; polyarthritis; combination therapy; biologic agents; TNF antagonists; infliximab
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infliximab plus Methotrexate (Experimental): infliximab 3-5 mg/kg every 6 weeks, plus methotrexate 15 mg/m2 weekly given orally (dose escalation if ACR Pedi less than 75). no oral prednisolone. intra-articular steroids allowed.
  Interventions: Drug: Infliximab plus methotrexate
- Combination of DMARDs (Experimental): methotrexate 15mg/m2 weekly given orally (dose escalation and parenteral injection if ACR Pedi less than 75), plus standard doses of sulfasalazine and hydroxychloroquine. no oral prednisolone. intra-articular steroids allowed.
  Interventions: Drug: Combination of DMARDs
- Methotrexate alone (Active Comparator): Conventional drug therapy: methotrexate 15mg/m2 weekly given orally (dose escalation and parenteral injection if ACR Pedi less than 75). no oral prednisolone. intra-articular steroids allowed.
  Interventions: Drug: Methotrexate alone

INTERVENTIONS:
Drug: Infliximab plus methotrexate — IFX given 3-5mg/kg every 6 weeks, oral MTX given 15mg/m2 weekly. If ACR Pedi 75 is not reached by week 12, MTX dose is doubled up to parenteral 30 mg/m2 weekly dose. If patient does not reach ACR Pedi 30 after dose escalation, failure.
  Other Names: IFX: Remicade, MTX: Trexan or Methotrexate
  Arms: Infliximab plus Methotrexate
Drug: Combination of DMARDs — IFX given 3-5mg/kg every 6 weeks, oral MTX given 15mg/m2 weekly, SSZ 40mg/kg up to 2000mg daily, HCQ 5mg/kg daily. If ACR Pedi 75 is not reached by week 12, MTX dose is doubled up to parenteral 30 mg/m2 weekly dose. If patient does not reach ACR Pedi 30 after dose escalation, failure.
  Other Names: MTX: Trexan or Methotrexate, SSZ: Salazopyrin, HCQ: Oxiklorin
  Arms: Combination of DMARDs
Drug: Methotrexate alone — Oral MTX given 15mg/m2 weekly. If ACR Pedi 75 is not reached by week 12, MTX dose is doubled up to parenteral 30 mg/m2 weekly dose. If patient does not reach ACR Pedi 30 after dose escalation, failure.
  Other Names: MTX: Trexan or Methotrexate
  Arms: Methotrexate alone

SUMMARY:
The objective of this study is to compare in very early polyarticular juvenile idiopathic arthritis (JIA) the efficacy, safety, and cost-benefit-ratio of three treatment strategies: biologic combination, combination of conventional disease-modifying drugs (DMARDs), and methotrexate alone.

DETAILED DESCRIPTION:
DMARD-naive polyarticular JIA patients with an early disease (onset less than 6 months) are randomized into one of three treatment strategies: (1) biological combination, i.e., anti-TNF therapy with infliximab plus methotrexate; (2) Combination of DMARDs with methotrexate, sulfasalazine, plus hydroxychloroquine; and (3) Methotrexate alone.

The efficacy is evaluated by American College of Rheumatology Pediatric (ACR Pedi) criteria based on 6 core set variables (CSVs): 1. no of active joints; 2. no. of joints with pain or tenderness and limitation of motion; 3. ESR (mm/hr); 4. the Childhood Health Assessment Questionnaire (CHAQ); 5. Physician's Visual Analogue Scale (VAS); 6. Patient/Parent VAS. To fulfill ACR Pedi 75 criteria, 3/6 CSVs have to improve 75% and not more than 1/6 CSV worsen more than 30%. All direct and indirect costs are documented.

The first phase of the study is open-label clinical trial lasting for 54 weeks. In the second phase of the study the patients are followed up to 5 years, and the long-term outcome of early aggressive therapy is analyzed. Serum, urine, and saliva samples are collected at 3 and 5 years for translational research.

ELIGIBILITY:
Inclusion Criteria:

* juvenile idiopathic arthritis
* arthritis lasting for at least 6 weeks but not more than 6 months
* polyarticular disease with at least 5 active joints with at least 3 joints with pain or tenderness and limitation of motion
* no previous treatment with DMARDs

Exclusion Criteria:

* systemic JIA
* any abnormality in the hematopoietic or lymphatic system
* any major concurrent medical condition
* inadequate psychosocial situation
* pregnancy
* a non-abstinent female with reproductive capacity without regular contraceptive use

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2003-05; Primary Completion 2007-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ACR Pedi 75 response | 54 weeks from baseline (0)

SECONDARY OUTCOMES:
clinically inactive disease | at 54 weeks
time spent in inactive disease | 0 to 54 weeks
time spent in ACR Pedi 75 | 0 to 54 weeks
Other ACR Pedi responses (30, 50, 70, 90, 100) | 0 to 54 weeks
drug survival | 54 weeks
occurrence of side-effects and adverse events | 0 to 54 weeks
cost-benefit ratio in each treatment arm | 0 to 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Lahdenne, MD, PhD, Study Director — Hospital for Children and Adolescents in Helsinki University Central Hospital
Locations (6):
- Finland (6):
  - Rheumatism Foundation Hospital, Heinola
  - Hospital for Children and Adolescents, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Central Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Background] Lahdenne P, Vahasalo P, Honkanen V. Infliximab or etanercept in the treatment of children with refractory juvenile idiopathic arthritis: an open label study. Ann Rheum Dis. 2003 Mar;62(3):245-7. doi: 10.1136/ard.62.3.245. PMID 12594111
- [Result] Tynjala P, Vahasalo P, Tarkiainen M, Kroger L, Aalto K, Malin M, Putto-Laurila A, Honkanen V, Lahdenne P. Aggressive combination drug therapy in very early polyarticular juvenile idiopathic arthritis (ACUTE-JIA): a multicentre randomised open-label clinical trial. Ann Rheum Dis. 2011 Sep;70(9):1605-12. doi: 10.1136/ard.2010.143347. Epub 2011 May 28. PMID 21623000
- [Derived] Tarkiainen M, Tynjala P, Vahasalo P, Aalto K, Kroger L, Rebane K, Lahdenne P, Martikainen J. Economic evaluation of infliximab, synthetic triple therapy and methotrexate in the treatment of newly diagnosed juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2022 Nov 16;20(1):97. doi: 10.1186/s12969-022-00748-w. PMID 36384562
- [Derived] Tarkiainen M, Tynjala P, Vahasalo P, Kroger L, Aalto K, Lahdenne P. Health-related quality of life during early aggressive treatment in patients with polyarticular juvenile idiopathic arthritis: results from randomized controlled trial. Pediatr Rheumatol Online J. 2019 Dec 16;17(1):80. doi: 10.1186/s12969-019-0370-1. PMID 31842940